CLINICAL TRIAL: NCT00173602
Title: The Burden of Peripheral Artery Occlusion Disease and Associated Factors in Peritoneal Dialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700811
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2005-08

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peritoneal Dialysis
MeSH Terms: conditions — Peripheral Vascular Diseases

SUMMARY:
The investigators want to evaluate the burden of peripheral artery occlusion disease in Taiwan peritoneal dialysis (PD) patients by using ankle-brachial pressure index (ABI) and toe-brachial pressure index (TBI). Furthermore, the investigators hope to demonstrate the possible casual factors of peripheral artery occlusion disease (PAOD) in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Receive stable peritoneal dialysis patients for more than 3 months

Exclusion Criteria:

* Active infection, malignancy and recent hospitalization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-09; Study Completion 2007-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Kang Chiang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan